CLINICAL TRIAL: NCT06168123
Title: Future Optimal Research and Care Evaluation - Aortic Stenosis
Acronym: FORCE-AoS
Status: Recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Clinical Professor, St. Antonius Hospital
Other Study IDs: Z23.069
Record Dates: First submitted 2023-10-20; First posted 2023-12-13 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-12

CONDITIONS: Severe Aortic Valve Stenosis; Moderate Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Quality of life questionnaires will be assessed in addition to standard care — Quality of life questionnaires will be assessed in addition to standard care

SUMMARY:
In the past decade the treatment of aortic valve stenosis has rapidly changed. At first, transcatheter aortic valve implantation (TAVI) was a last resort option for inoperable patients. Nowadays, it more and more becomes an alternative to surgical aortic valve replacement (SAVR) - also in younger and lower risk patients. This poses important questions to clinical practise regarding the optimal life-time management of each individual patient. Which involves (durability of) treatment modality (surgical vs. transcatheter vs. conservative treatment) as well as the duration and type of the required antithrombotic treatment.

Objective: to evaluate the effect of treatment modality (surgical vs. transcatheter vs. conservative treatment) and its complications on quality of life and survival in AoS patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Severe or moderate aortic stenosis

No exclusion criteria are applicable to this registry

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe or moderate aortic stenosis
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life as assessed by the EQ-5D-5L | Until completion of the study (August 1, 2027)
  The EQ-5D-5L is a standardized health-related quality of life instrument that assesses individuals across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It generates a health profile that can be converted into a single index value, commonly ranging from -0.594 to 1, where 1 represents full health, 0 indicates a state equivalent to death, and negative values reflect health states perceived as worse than death.
Quality of life as assessed by the KCCQ | Until completion of the study (August 1, 2027)
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific instrument assessing heart failure patients across domains such as Total Symptoms, Physical Limitation, and Quality of Life, with scores ranging from 0 to 100. Higher scores indicate better health-related quality of life, while lower scores suggest increased symptomatology and functional limitations in heart failure patients.
Quality of life as assessed by the SF-12 | Until completion of the study (August 1, 2027)
  The Short Form 12 (SF-12) is a widely used health survey that measures health-related quality of life across physical and mental domains. It generates two summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS), both ranging from 0 to 100, where higher scores indicate better health status, and these summaries provide a concise assessment of an individual's overall physical and mental well-being.

SECONDARY OUTCOMES:
Mortality according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Neurological events according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Hospitalisation according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Bleeding and transfusions according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Vascular and access-related complications according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Cardiac structural complications according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Other procedural or valve-related complications according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
New conduction disturbances and arrhythmias according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Acute kidney injury according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Myocardial infarction according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Bioprosthetic valve dysfunction according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Leaflet thickening and reduced motion according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Clinically significant valve thrombosis according the VARC-3 criteria | Until completion of the study (August 1, 2027)
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided